CLINICAL TRIAL: NCT07107009
Title: Climate Change and Air Contamination: Artificial Intelligence Applied on the Correlation Between Air Pollutants and Non-communicable Respiratory Diseases in Europe (ClimAIr)
Brief Title: ClimAIr: AI to Assess the Impact of Pollution and Climate on Respiratory Health in Europe
Acronym: ClimAIr
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Theramed Healthcare SRL (Romania) (Unknown); Centre Hospitalier Universitaire de Toulouse, FRANCE (Unknown); Charite-Universitaetsmedizin Berlin (Germany) (Unknown); Aristotelio Panepistimio Thessalonikis (Greece) (Unknown); Uniwersytet Medyczny w Lodzi (Poland) (Unknown); Universita degli Studi di Milano (Italy) (Unknown); Bukovinian State Medical University (Ukraine) (Unknown); Luxembourg Institute of Health (Luxembourg) (Unknown); Andaluz Health Service (Other Government)
Responsible Party: Sponsor
Other Study IDs: 101156799-2 ClimAIr
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: Air contamination; Air pollutants; Non-communicable respiratory diseases; Climate change; ClimAIr
MeSH Terms: conditions — Rhinitis, Allergic; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Peripheral blood : for serum ,DNA isolation and cellular assays. Nasal lavage: Bilateral lavage using isotonic saline by Naclerio method. Skin tape strips: 16 consecutive D-Squame tape strips applied to forearm for skin tissue sampling.
  Analyses performed on samples include:
  Proteomics (Olink®) on serum and nasal lavage supernatant Targeted metabolomics (LC-MS and GC-MS) on serum and nasal lavage DNA methylation profiling (Illumina EPIC array) from PBMC DNA Flow cytometry of PBMC cultured with pollen to assess lymphocyte proliferation and antibody production Multiplex ELISA for cytokine quantification in PBMC culture supernatants Microbiota analysis (16S, 18S, ITS2 sequencing) from nasal lavage pellets and skin tape strips
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- P01 - General Exposure Cohort: >200 AR patients per environmental condition. Includes patients exposed to various air pollutants, aiming to detect deleterious clinical effects.
- P02 - Omics Synergistic Subgroup: Subgroup of 20 patients per environmental condition from P01. Selected based on exposure to multiple pollutants with observed synergistic effects on omics parameters.
- S01 - Allergen-Specific Immune Response Subgroup: Subgroup of 25 patients per pollution condition from P01. Selected for in vitro assays to evaluate proliferation of peripheral allergen-specific lymphocytes in response to polluted pollen exposure.

SUMMARY:
The ClimAIr project will expand the evidence-based understanding of climate change, air pollution, and non-communicable respiratory diseases by using Artificial Intelligence (AI) tools. It will gather data on greenhouse gases levels and disaster risks, information on serious air pollutants and respiratory diseases' prevalence. The AI powered tools will be employed to generate better intervention methods and improve public health outcomes.

Federated Learning (FL) will be used to develop AI models to protect patients' privacy. By raising public awareness and delivering the ClimAIr tool - specifically designed to health workers, urban planners and policy makers - the project aims to influence policy decisions, promote healthier environments, and reduce respiratory diseases in Europe, which will be tested and validated the ClimAIr tool in specific municipalities that are part of the project. ClimAIr draws on a consortium of 21 partners from 15 European countries, including carefully selected health centres across Europe - in Spain, Luxembourg, Ukraine, Italy, France, Germany, Greece, Romania and Poland - focused on respiratory diseases, which will provide disease data and explore metabolic routes of the studied contaminants/diseases. ClimAIr is composed of an interdisciplinary team formed by research centres, ethical AI and modelling experts, SSH specialists, municipal governance, and a Communication & Dissemination (C&D) expert team dedicated to achieving and spread the results of the project.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with health insurance based in Malaga, Milan, Luxembourg, Thessalonikki, Lodz, Berlin, Toulousse, Chervnivtsi and Brasov (the places where environmental/climate information will be obtained from, only one recruitment place for partner).
2. 3-year history of chronic rhinitis symptoms during the corresponding pollen season, while residing in the same household AND attending the same school/college or holding the same job position.
3. Positive SPT and serum allergen-specific IgE >0.35 kUA/L. The pollen species driving the nasal symptoms will be Olea europaea, Phleum pratense or Betula pendula.
4. Patients can be sensitized to other aeroallergens if the nasal symptoms occur exclusively or aggravate unequivocally during the pollen season of the three allergens of interest.

Exclusion Criteria:

Lack of reliable information in e-health records, allergen immunotherapy (any allergen) during the previous 5 years, systemic immunosuppressants or biologicals in the previous six months, chronic rhinosinusitis, and severe systemic conditions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pacients with 3-year history of chronic rhinitis symptoms during the corresponding pollen seasonp ositive SPT and serum allergen-specific IgE >0.35 kUA/L.
Sampling Method: Non-Probability Sample
Enrollment: 1906 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean Symptom Score of Allergic Rhinitis Patients by Environmental Exposure | Retrospective data collected over a 3-year period prior to study enrollment.
  Mean allergic rhinitis symptom scores retrieved from electronic health records (EHR), stratified by environmental exposure levels (pollutants and climate factors), using the Observational Medical Outcomes Partnership (OMOP) common data model.
Proteomic Biomarker Levels (NPX) by Environmental Exposure | Samples collected prospectively between months 10 and 15 (October-March, out-of-pollen season).
  Proteomic profiles measured using Olink® assays in serum and nasal lavage of allergic rhinitis patients, stratified by environmental exposure.

SECONDARY OUTCOMES:
SO1: Effect of air pollution on adaptive immune responses to allergenic pollen | Sample collection and analysis performed prospectively between months 10 and 24.
  Evaluation of the immune response of peripheral blood mononuclear cells (PBMCs) from allergic rhinitis patients exposed to different environmental conditions, after in vitro stimulation with pollen samples previously exposed to varying pollution levels. The response will be characterized by proliferation of allergen-specific lymphocyte subsets and cytokine production.
SO1: Proliferative responses of allergen-specific lymphocytes to pollen exposed to pollution | Assays conducted on samples collected between months 10 and 24.
  Measurement of lymphocyte proliferation using CFSE-labeled PBMCs incubated with pollen (Olea europaea, Phleum pratense, Betula pendula) grown under different pollution conditions.
SO1: Cytokine release from allergen-specific lymphocytes in response to polluted pollen | Analysis performed between months 10 and 24, post-sample collection.
  Quantification of cytokines released in the supernatants of PBMC cultures stimulated with pollen under different pollution conditions. A multiplex ELISA panel will be used to measure Th1, Th2, Th9, and regulatory cytokine

IPD SHARING:
Plan to Share IPD: Undecided